CLINICAL TRIAL: NCT07345039
Title: Comparison of Infraorbital-Infratrochlear Nerve Block and Transnasal Sphenopalatine Ganglion Block on Postoperative Analgesia and Recovery Outcomes in Septorhinoplasty: A Prospective, Randomized, Double-Blind Clinical Trial
Brief Title: Infraorbital-Infratrochlear Block vs Sphenopalatine Ganglion Block for Postoperative Analgesia in Septorhinoplasty.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12.2.2025-521
Record Dates: First submitted 2025-12-10; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, randomized and double-blind clinical trial comparing infraorbital-infratrochlear nerve block with transnasal sphenopalatine ganglion block in patients undergoing septorhinoplasty.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, surgeons, anesthesiologists assessing postoperative outcomes, follow-up investigators, and data analysts were all blinded to group allocation throughout the perioperative period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infraorbital-Infratrochlear Nerve Block (ION-ITN Block) (Active Comparator): Infraorbital-Infratrochlear Nerve Block (ION-ITN Block)
  Interventions: Procedure: Infraorbital-Infratrochlear Nerve Block
- Sphenopalatine Ganglion Block (Active Comparator): Transnasal Sphenopalatine Ganglion Block (SPG Block)
  Interventions: Procedure: Transnasal Sphenopalatine Ganglion Block

INTERVENTIONS:
Procedure: Infraorbital-Infratrochlear Nerve Block — Bilateral infraorbital and infratrochlear nerve block performed with 0.5% bupivacaine after induction of general anesthesia
  Arms: Infraorbital-Infratrochlear Nerve Block (ION-ITN Block)
Procedure: Transnasal Sphenopalatine Ganglion Block — Transnasal sphenopalatine ganglion block performed after induction of general anesthesia using local anesthetic-soaked applicators
  Arms: Sphenopalatine Ganglion Block

SUMMARY:
This prospective, randomized, double-blind clinical trial aims to compare the postoperative analgesic efficacy and recovery outcomes of infraorbital-infratrochlear nerve block and transnasal sphenopalatine ganglion block in patients undergoing septorhinoplasty under general anesthesia. Adult patients aged 18-65 years with ASA I-II status will be randomized to receive either bilateral infraorbital-infratrochlear block or transnasal sphenopalatine ganglion block after induction of anesthesia. Postoperative outcomes including pain scores (NRS at 0-2 h, 2-8 h, and 8-24 h), emergence agitation, Riker Sedation-Agitation Scale (RSAS) scores, time to first rescue analgesic, total tramadol consumption, adverse events, surgical site complications, and patient satisfaction will be assessed and compared between groups.

DETAILED DESCRIPTION:
This study is designed to evaluate the postoperative analgesic efficacy and clinical outcomes of two regional anesthesia techniques-infraorbital-infratrochlear nerve block (ION-ITN block) and transnasal sphenopalatine ganglion block (usg guided sphenopalatine ganglion block,SPG block)-in patients undergoing septorhinoplasty under general anesthesia. Eligible patients aged 18-65 years with ASA physical status I-II will be randomly assigned to one of two intervention groups. Blocks will be performed after induction by an anesthesiologist not involved in postoperative assessment. Patients, surgeons, anesthesiologists performing postoperative evaluations, follow-up investigators, and data analysts will remain blinded to group allocation.

Postoperative outcomes will include pain intensity assessed using the Numerical Rating Scale (NRS) at 0-2, 2-8, and 8-24 hours after surgery, agitation between extubation and PACU discharge assessed with the Riker Sedation-Agitation Scale (RSAS), emergence agitation (RSAS ≥5), time to first rescue analgesic, and total tramadol consumption within 24 hours. Additional outcomes include postoperative nausea and vomiting, cardiovascular and respiratory adverse events, surgical site complications (edema, hematoma, neurologic deficit), and patient satisfaction measured by a 5-point Likert scale. Preoperative demographics, BMI, ASA class, comorbidities, anesthesia and surgery duration, and intraoperative remifentanil consumption will be recorded. The study aims to determine whether SPG block provides superior postoperative analgesia compared with ION-ITN block in septorhinoplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years.
* Scheduled for septorhinoplasty under general anesthesia.
* American Society of Anesthesiologists (ASA) Physical Status I-II.
* Ability to cooperate with postoperative evaluations.
* Provision of written informed consent.

Exclusion Criteria:

* Allergy or contraindication to local anesthetics used in the study.
* Coagulopathy or anticoagulant therapy.
* Local infection at the nerve block application sites.
* Severe nasal anatomical abnormalities preventing transnasal block application.
* Psychiatric disorders affecting pain or agitation assessment..
* Chronic pain conditions or chronic opioid use.
* Neurological disorders affecting sensory perception.
* Refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 0-24 hours postoperative
  Pain intensity assessed using the Numerical Rating Scale (NRS, 0-10) at three postoperative intervals: 0-2 hours, 2-8 hours, and 8-24 hours. Higher scores indicate greater pain.
Postoperative Agitation | Immediate postoperative period (from extubation to discharge from the post-anesthesia care unit [PACU]; up to 2 hours)
  Agitation severity assessed using the Riker Sedation-Agitation Scale (RSAS). The highest postoperative RSAS score is recorded. RSAS ≥5 is defined as emergence agitation.

SECONDARY OUTCOMES:
Total Tramadol Consumption | First 24 hours postoperative
  Total amount of intravenous tramadol administered as postoperative analgesia.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-24 hours postoperative
  Occurrence of nausea or vomiting requiring treatment with ondansetron.
Adverse Events in PACU | Immediate postoperative period (from extubation to discharge from the post-anesthesia care unit [PACU]; up to 2 hours)
  Respiratory or cardiovascular events including oxygen desaturation, airway obstruction, hypotension, hypertension, or arrhythmia.
Patient Satisfaction Score | At 24 hours postoperative
  Patient satisfaction assessed using a 5-point Likert scale (1 = very unsatisfied, 5 = very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Can E, Akkaya OT. A Comparison of Transnasal Versus Ultrasound-Guided Suprazygomatic Approaches for Sphenopalatine Ganglion Blocks in Persistent Idiopathic Facial Pain. Ann Indian Acad Neurol. 2025 Mar 1;28(2):189-195. doi: 10.4103/aian.aian_713_24. Epub 2025 Mar 13. PMID 40087987